CLINICAL TRIAL: NCT06801015
Title: A Randomized, Placebo-Controlled Trial of the Effects of Long-Acting GLP-1 or Dual Incretin (GLP-1 and GIP) Modulation on Gastric Motor Functions
Brief Title: Effects of Long-Acting GLP-1 (Glucagon-like Peptide-1) or Dual Incretin (GLP-1 and GIP [Glucose-dependent Insulinotropic Peptide]) Modulation on Gastric Motor Functions
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-011786
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide; Tirzepatide

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of the effects of semaglutide, tirzepatide, and placebo with concealed allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Concealed allocation with masking of medications administered by subcutaneous injection once per week; blinding of all investigators since medication is dispensed by research pharmacy not by clinical research trials unit
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- semaglutide (Experimental): Administered by subcutaneous injection once per week in accordance with FDA approved escalation as well as maintenance treatment
  Interventions: Drug: Semaglutide
- Tirzepatide (Experimental): Administered by subcutaneous injection once per week in accordance with FDA approved escalation as well as maintenance treatment
  Interventions: Drug: Tirzepatide
- placebo (Placebo Comparator): Administered by subcutaneous injection once per week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Both interventions are approved by FDA for the treatment of obesity and are administered by subcutaneous injection once per week
  Arms: semaglutide
Drug: Tirzepatide — Both interventions are approved by FDA for the treatment of obesity and are administered by subcutaneous injection once per week
  Arms: Tirzepatide
Drug: Placebo — Placebo administered by subcutaneous injection once per week.
  Arms: placebo

SUMMARY:
The purpose of this study is to compare effects of weekly SQ semaglutide 2.4mg SQ, SQ tirzepatide 10mg, and placebo administered for 24 weeks on GES measured repeatedly at baseline, 16 weeks, 24 weeks, 28 weeks, 4 weeks after stopping the medication, and accommodation and satiation at 24 weeks compared to baseline.

ELIGIBILITY:
PLEASE NOTE: Potential participants must reside within 50 miles of Mayo Clinic for 7 consecutive months due to non-mobile GI imaging cameras.

Inclusion criteria:

* Adults (18-75 years) who have BMI >30 or >27kg/m2 who also have prediabetes or T2DM on diet treatment only
* Able to reside within 50 miles of Mayo Clinic for the duration of the study
* Not currently on treatment (exceptions below) for cardiac, pulmonary, GI, hepatic, renal, hematological, neurological, or endocrine disorders.
* Biological sex: men or women. We shall attempt to recruit equal proportions of men and women. Women of childbearing potential will be using an effective form of contraception and have negative pregnancy tests within 48 hours of enrollment and before each isotope-based radiation exposure as part of the tests for gastric emptying. In addition, monthly urine pregnancy tests will be performed in females with childbearing potential.

Exclusion criteria:

* Weight exceeding 137kg (safety limit of camera for measuring gastric volumes)
* Abdominal surgery other than appendectomy, Caesarian section or tubal ligation, cholecystectomy
* Chronic GI diseases, systemic disease or medications that could affect GI motility, appetite or absorption
* Patients with a personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia II
* Patients with T2DM on GLP-1RAs, amylin agonists/analogs (e.g. pramlintide), insulin, sulfonylureas (all due to risk of hypoglycemia with semaglutide or tirzepatide treatment); or on metformin, acarbose or DPP-4 inhibitors (e.g. sitagliptin and vildagliptin).
* Past or current history of pancreatitis, gallstones, history of alcoholism, blood triglyceride levels > 500mg/dL
* Significant untreated psychiatric dysfunction or an active eating disorder (Clark et al 2007, Cunningham et al 2012) based on screening with the Hospital Anxiety and Depression Inventory [HAD (Zigmond & Snaith 1983)], a self-administered alcoholism screening test [AUDIT-C (Bush et al 1998)], and the Questionnaire on Eating and Weight Patterns-Revised [binge eating disorders and bulimia (Yanovski et al 2015)]. If such a dysfunction is identified by a HAD score >11 on either the anxiety or depression subscales or difficulties with substance or eating disorders, the participant will be interviewed by a study investigator and, if excluded, will be given a referral letter to his/her primary care doctor for further appraisal and follow-up treatment.
* Intake of any medication (except multivitamins) within 7 days of the study. Exceptions are birth control pill, estrogen and thyroxine replacement, and medication administered for co-morbidities as long as they do not alter gastric functions. Thus, statins for hyperlipidemia, diuretics, β-adrenergic blockers, ACE inhibitors and angiotensin antagonists for hypertension are permissible. In contrast, resin sequestrants for hyperlipidemia (Psichas et al 2012), α2-adrenergic agonists for hypertension, are not permissible due to effects on stomach or appetite.
* Documented delayed gastric emptying: gastric emptying T1/2 >174 min or gastric retention at 4 hours >25% based on 5-95%ile of 319 controls' GES of the same meal (320kcal, 30% fat) (Camilleri et al 2012a, Table 1)
* Hypersensitivity to semaglutide or tirzepatide
* Participate in highly intense physical activity program that could potentially interfere with study interpretation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying of solids T1/2 min, that is time for half meal to empty from stomach | Measurement at baseline, after 16 and 24 weeks' treatment, and at 28 weeks (off treatment for 4 weeks)
  Gastric emptying of an egg meal measured by scintigraphy
Body weight | Measurement at baseline, after 16 and 24 weeks' treatment, and at 28 weeks (off treatment for 4 weeks)
  Measurement of body weight using weight scales

SECONDARY OUTCOMES:
Calories to fullness, kilocalories (kcal) | Measurement at baseline, and after 24 weeks' treatment
  Measurement of kilocalorie intake at comfortable fullness based on Ensure liquid nutrient
Maximum tolerated calories, kilocalories (kcal) | Measurement at baseline, and after 24 weeks' treatment
  Measurement of kilocalorie intake at maximal fullness based on Ensure liquid nutrient
Fasting gastric volume, milliliters (mL) | Measurement at baseline, and after 24 weeks' treatment
  Measurement of gastric volume during fasting using 99mTc-SPECT (single photon emission computed tomography) imaging
Gastric accommodation vol (postprandial minus fasting volume), milliliters (mL) | Measurement at baseline, and after 24 weeks' treatment
  Measurement of gastric volume following 300 mL of Ensure using 99mTc-SPECT (single photon emission computed tomography) imaging
Peak postprandial GLP-1 (glucagon-like peptide-1) pmol/L | Measurement at baseline, and after 24 weeks' treatment
  GLP-1 measured fasting, and 15, 45, and 90 minutes postprandially
Peak postprandial peptide tyrosine tyrosine (PYY) pmol/L | Measurement at baseline, and after 24 weeks' treatment
  PYY measured fasting, and 15, 45, and 90 minutes postprandially
DEXA (dual energy X-ray absorptiometry) body composition | Measurement at baseline, and after 24 weeks' treatment
  Body composition (including total body fat) by dual-energy X-ray absorptiometry (DEXA) technology

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No